CLINICAL TRIAL: NCT01723228
Title: A 24-Week, Multicenter, Randomized, Double-blind, Placebo-Controlled, Add-on, Parallel-Group Study to Assess the Effect of Rasagiline on Cognition in Patients With Parkinson's Disease
Brief Title: Parallel-Group Study to Assess the Effect of Rasagiline on Cognition in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVP-1012/PM106
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Cognition; Rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Mesylates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline 1.0 mg/day (Experimental): Rasagiline 1 mg oral tablets once daily for 24 weeks
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): Placebo oral tablets once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline
  Other Names: Azilect® (rasagiline [N-propargyl-1-(R)-aminoindan] mesylate); TVP-1012
  Arms: Rasagiline 1.0 mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 24-week, multicenter, randomized, double-blind, placebo-controlled, add-on, parallel-group study to evaluate the effect of rasagiline on cognitive function in adults with mild cognitive impairment (MCI) in Parkinson's disease (PD-MCI).

ELIGIBILITY:
Inclusion Criteria:

1. Nondemented man or woman 45 through 80 years of age with idiopathic Parkinson's disease (PD) based on the United Kingdom (UK) Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
2. Hoehn and Yahr stage ≥ 1 (symptoms on only 1 side of the body) with treatment and ≤ 3 (mild-to-moderate bilateral disease; some postural instability; physically independent)
3. Mild cognitive impairment in Parkinson's disease based on the Movement Disorder Society (MDS) Task Force Diagnostic Criteria and the Montreal Cognitive Assessment (MoCA) rating scale (range, 20-25, inclusive)
4. Medically stable outpatient, based on the investigator's judgment
5. The patient is on a stable dopaminergic medication regimen for ≥ 30 days before entering the study (Screening/Baseline Visit)
6. Other inclusion criteria apply; please contact the site for more information

Exclusion Criteria:

1. Clinically relevant history of vascular disease (eg, stroke)
2. History of melanoma
3. History of deep brain stimulation (DBS)
4. Impaired hepatic function, based on the investigator's judgment
5. Psychosis or is receiving antipsychotic treatment
6. Clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation, based on the investigator's judgment
7. Other exclusion criteria apply; please contact the site for more information

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (40):
- United States (40):
  - Teva Investigational Site 036, Birmingham, Alabama
  - Teva Investigational Site 047, Sun City, Arizona
  - Teva Investigational Site 004, Irvine, California
  - Teva Investigational Site 016, La Jolla, California
  - Teva Investigational Site 042, Long Beach, California
  - Teva Investigational Site 041, San Bernardino, California
  - Teva Investigational Site 048, Denver, Colorado
  - Teva Investigational Site 038, Englewood, Colorado
  - Teva Investigational Site 035, Danbury, Connecticut
  - Teva Investigational Site 034, Manchester, Connecticut
  - Teva Investigational Site 037, New London, Connecticut
  - Teva Investigational Site 026, Washington D.C., District of Columbia
  - Teva Investigational Site 015, Boca Raton, Florida
  - Teva Investigational Site 021, Jacksonville, Florida
  - Teva Investigational Site 033, Ormond Beach, Florida
  - Teva Investigational Site 020, Port Charlotte, Florida
  - Teva Investigational Site 017, St. Petersburg, Florida
  - Teva Investigational Site 019, Atlanta, Georgia
  - Teva Investigational Site 003, Chicago, Illinois
  - Teva Investigational Site 006, Chicago, Illinois
  - Teva Investigational Site 008, Chicago, Illinois
  - Teva Investigational Site 025, Kansas City, Kansas
  - Teva Investigational Site 009, Lexington, Kentucky
  - Teva Investigational Site 046, Baton Rouge, Louisiana
  - Teva Investigational Site 024, Boston, Massachusetts
  - Teva Investigational Site 031, Las Vegas, Nevada
  - Teva Investigational Site 030, New Brunswick, New Jersey
  - Teva Investigational Site 014, Albany, New York
  - Teva Investigational Site 045, Commack, New York
  - Teva Investigational Site 013, Kingston, New York
  - Teva Investigational Site 010, New York, New York
  - Teva Investigational Site 040, New York, New York
  - Teva Investigational Site 022, Asheville, North Carolina
  - Teva Investigational Site 005, Raleigh, North Carolina
  - Teva Investigational Site 018, Toledo, Ohio
  - Teva Investigational Site 028, Philadelphia, Pennsylvania
  - Teva Investigational Site 012, Nashville, Tennessee
  - Teva Investigational Site 002, San Antonio, Texas
  - Teva Investigational Site 011, Salt Lake City, Utah
  - Teva Investigational Site 001, La Crosse, Wisconsin

REFERENCES:
- [Background] Hanagasi HA, Gurvit H, Unsalan P, Horozoglu H, Tuncer N, Feyzioglu A, Gunal DI, Yener GG, Cakmur R, Sahin HA, Emre M. The effects of rasagiline on cognitive deficits in Parkinson's disease patients without dementia: a randomized, double-blind, placebo-controlled, multicenter study. Mov Disord. 2011 Aug 15;26(10):1851-8. doi: 10.1002/mds.23738. Epub 2011 Apr 15. PMID 21500280

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Started | 86 | 84
Completed | 78 | 73
Not Completed | 8 | 11
Not completed — Adverse Event | 2 | 6
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline 1.0 mg/Day | Placebo | Total
Number analyzed (Participants) | 86 | 84 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (7.44) | 68.1 (8.22) | 67.5 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 65 | 68 | 133

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 24 in the Scales for Outcomes in Parkinson's Disease-Cognition (SCOPA-COG) Summary Score
Description: The SCOPA-COG consists of evaluations in 4 domains: memory, attention, executive functioning, and visuospatial functioning.Scores range from 0 to 43, with higher scores reflecting better performance.
Time Frame: Baseline to Week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline SCOPA-COG assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | 1.6 (0.45) | 0.8 (0.47)
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.2204, repeated measures model; The statistical model is a repeated measures model with visit by treatment interaction, center, baseline score, and age as fixed effects; Least Squares Mean Difference = 0.8, 95% CI 2-sided [-0.48 to 2.05]

2. Secondary Outcome: Change From Baseline to Week 24 in the Montreal Cognitive Assessment (MoCA) Score
Description: The MoCA assesses 8 cognitive areas: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. Scores range from 0 (worst) to 30 (best).
Time Frame: Baseline to Week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline MoCA assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | 0.9 (0.32) | 1.0 (0.34)
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.8428, Repeated Measures Model; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.99 to 0.81]

3. Secondary Outcome: Change From Baseline to Week 24 in the Penn Daily Activities Questionnaire (PDAQ) Score
Description: The PDAQ is a 15-item questionnaire that assesses the patient's difficulty with activities of daily living. The total score has a range of 0 (no impairment) to 60 (severe impairment).
Time Frame: Baseline to Week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline PDAQ assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -0.9 (0.72) | -0.1 (0.75)
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.4796, ANCOVA; The statistical model is an analysis of covariance (ANCOVA) with treatment, center, baseline score, and age as fixed effects; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.74 to 1.30]

4. Secondary Outcome: Alzheimer's Disease Cooperative Study's Clinical Global Impression of Change Modified for Mild Cognitive Impairment (ADCS MCI-CGIC) Score at Week 24
Description: The ADCS MCI-CGIC score is generated in the context of a semi-structured interview and is an indication of the change in the participant's global status, cognition, behavior, and functional abilities (FA) on a 7-point scale, with the best score being 'marked improvement' and the worst being 'marked worsening.'
Time Frame: Week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline ADCS MCI-CGIC assessment. n=number of participants with the given assessment.
Measure: Number; unit: participants
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 80 | 82
participants
  CGIC: Marked improvement; n=78, 79 | 1 | 4
  CGIC: Moderate improvement; n=78, 79 | 9 | 7
  CGIC: Minimal improvement; n=78, 79 | 11 | 23
  CGIC: No change; n=78, 79 | 42 | 33
  CGIC: Minimal worsening; n=78, 79 | 14 | 12
  CGIC: Moderate worsening; n=78, 79 | 1 | 0
  CGIC: Marked worsening; n=78, 79 | 0 | 0
  CGIC Cognition: Marked improvement; n=77, 79 | 0 | 3
  CGIC Cognition: Moderate improvement; n=77, 79 | 9 | 4
  CGIC Cognition: Minimal improvement; n=77, 79 | 15 | 18
  CGIC Cognition: No change; n=77, 79 | 41 | 44
  CGIC Cognition: Minimal worsening; n=77, 79 | 9 | 8
  CGIC Cognition: Moderate worsening; n=77, 79 | 3 | 2
  CGIC Cognition: Marked worsening; n=77, 79 | 0 | 0
  CGIC Behavior: Marked improvement; n=76, 79 | 0 | 3
  CGIC Behavior: Moderate improvement; n=76, 79 | 4 | 1
  CGIC Behavior: Minimal improvement; n=76, 79 | 11 | 11
  CGIC Behavior: No change; n=76, 79 | 54 | 62
  CGIC Behavior: Minimal worsening; n=76, 79 | 7 | 2
  CGIC Behavior: Moderate worsening; n=76, 79 | 0 | 0
  CGIC Behavior: Marked worsening; n=76, 79 | 0 | 0
  CGIC FA: Marked improvement; n=76, 79 | 0 | 3
  CGIC FA: Moderate improvement; n=76, 79 | 5 | 4
  CGIC FA: Minimal improvement; n=76, 79 | 13 | 12
  CGIC FA: No change; n=76, 79 | 44 | 55
  CGIC FA: Minimal worsening; n=76, 79 | 12 | 5
  CGIC FA: Moderate worsening; n=76, 79 | 2 | 0
  CGIC FA: Marked worsening; n=76, 79 | 0 | 0
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC; Test type: Superiority or Other; p = 0.1148, Proportional Odds Model; The statistical model is a proportional odds model with terms for treatment, center, and age; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.89 to 2.93]
Statistical Analysis 2: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC; Test type: Superiority or Other; p = 0.1052, Cochran-Mantel-Haenszel; For the Cochran-Mantel-Haenszel (CMH) p-value, the statistical model is a CMH test controlling for center with scores=modridit option
Statistical Analysis 3: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Cognition; Test type: Superiority or Other; p = 0.8857, Proportional Odds Model; The statistical model is a proportional odds model with terms for treatment, center, and age; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.52 to 1.75]
Statistical Analysis 4: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Cognition; Test type: Superiority or Other; p = 0.9945, Cochran-Mantel-Haenszel — For the CMH p-value, the statistical model is a CMH test controlling for center with scores=modridit option
Statistical Analysis 5: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Behavior; Test type: Superiority or Other; p = 0.6909, Proportional Odds Model; The statistical model is a proportional odds model with terms for treatment, center, and age; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.56 to 2.43]
Statistical Analysis 6: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Behavior; Test type: Superiority or Other; p = 0.6639, Cochran-Mantel-Haenszel; For the CMH p-value, the statistical model is a CMH test controlling for center with scores=modridit option
Statistical Analysis 7: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Functional Abilities; Test type: Superiority or Other; p = 0.3204, Proportional Odds Model; The statistical model is a proportional odds model with terms for treatment, center, and age; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.72 to 2.68]
Statistical Analysis 8: Comparison: Rasagiline 1.0 mg/Day vs Placebo; CGIC Functional Abilities; Test type: Superiority or Other; p = 0.3331, Cochran-Mantel-Haenszel; For the CMH p-value, the statistical model is a CMH test controlling for center with scores=modridit option

5. Secondary Outcome: Change From Baseline to Week 24 in the Unified Parkinson's Disease Rating Scale (UPDRS), Motor Subscale (Part 3), Version 3, Score
Description: UPDRS Part 3 (motor examination subscale) comprises 14 items assessing the motor disabilities of the patient at the time of the visit. The participant's speech, facial expressions, ability to arise from a chair (with arms folded), posture, gait, postural stability (retropulsion test), and body bradykinesia and hypokinesia are assessed. In addition, the following evaluations require assessment of the face, neck or extremities: tremor at rest, action or postural tremor of hands, rigidity, finger taps, hand movements (open and close), rapid alternating movements of hands (pronation and supination), and leg agility (tap heel on ground). This evaluation is performed while the participant is in the 'on' phase. Each item is assessed on a scale from 0 (normal, absent, or none) to 4 (severe impairment), which are summed to get the sub-scale score. The total scale is 0-57 with a higher score indicating more severe symptoms; a decrease in the scores indicates improvement.
Time Frame: Baseline to Week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline UPDRS Motor Subscale (Part 3) assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 81 | 79
units on a scale | -3.7 (0.70) | -1.2 (0.73)
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0151, Repeated Measures Model; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-4.47 to -0.49]

6. Secondary Outcome: Change From Baseline to Week 24 in UPDRS, Activities of Daily Living (ADL) Subscale (Part 2), Version 3, Score
Description: UPDRS Part 2 (ADL subscale) comprises 13 items evaluating the impact of PD on patients' ADL (in both the on and off states) in the week prior to the visit. The following 13 ADL are assessed: speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed and adjusting bed clothes, falling (unrelated to freezing), freezing when walking, walking, tremor, and sensory complaints related to Parkinsonism. Each item is assessed on a scale from 0 (normal, absent, or none) to 4 (severe impairment), which are summed to get the sub-scale score. The total scale is 0-52 with a higher score indicating more severe symptoms; a decrease in the scores indicates improvement.
Time Frame: Baseline to week 24 (or early discontinuation)
Population: Modified intent-to-treat population: all participants who were randomized, received at least 1 dose of study drug and had at least 1 postbaseline UPDRS ADL Subscale (Part 2) assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -0.9 (0.43) | 1.4 (0.45)
Statistical Analysis 1: Comparison: Rasagiline 1.0 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0003, Repeated Measures Model; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-3.53 to -1.08]

ADVERSE EVENTS:
Time Frame: Baseline through Week 24
Arm/Group | Rasagiline 1.0 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/86 | 1/84
Other Adverse Events (participants affected / at risk) | 24/86 | 14/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline 1.0 mg/Day (N=86) | Placebo (N=84)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline 1.0 mg/Day (N=86) | Placebo (N=84)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.